CLINICAL TRIAL: NCT04789369
Title: The Relationship Between Fear of Movement, Functionality and Quality of Life in Elite Athletes With an Ankle Instability History
Brief Title: Fear of Movement, Functionality and Quality of Life in Elite Athletes With an Ankle Instability History
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özgül Öztürk, Assistant Professor, Acibadem University
Other Study IDs: 2020-04/14
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Ankle Sprains
Keywords: Quality of life; Fear of movement; Functionality; Ankle sprain
MeSH Terms: conditions — Ankle Injuries; Kinesiophobia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Questionnaires — Assessing the behavioral metrics (quality of life, functionality and fear of movement) with appropriate measurement tools

SUMMARY:
Ankle sprain is frequently experienced by individuals participating in different sports activities. Ankle sprains have been shown to result in a decrease in level of physical activity and persistence of some symptoms for a long time. In this case, it is predicted that ankle sprains may affect the quality of life as well as functionality. Also, ankle sprain history may result in increased fear of movement, which may delay return to sports. This study aimed to examine the relationship between foot and ankle functionality, fear of movement and quality of life of elite athletes with a history of ankle sprain.

ELIGIBILITY:
Inclusion Criteria:

* No injury to the upper or lower extremities during data collection,
* Being older than 18 years of age,
* Individuals who volunteer to participate.

Exclusion Criteria:

. Having had ankle surgery,

* Has had an injury to his lower extremity in the last 3 months,
* Individuals with a history of neurological / neuropsychiatric disease or arthritis will be excluded from the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Athletes who are participating in sportive activities regularly
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure | 1 day
  The Foot and Ankle Ability Measure will be used to determine the ankle functionality. This scale was developed to determine lower extremity functional level. It evaluates the level of difficulty of the person in activities in daily life in 21 items with a 5-point Likert-type scale, which means "4 = not difficult at all" and "0 = I cannot do it". At the same time, it can be reported within the scope of the scale that the specified activity cannot be implemented. High score means better functions.
Short Form-12 | 1 day
  Short-Form 12 is a valid and reliable scale for determining the level of quality of life. This scale consists of 12 items and can be scored as 8 subscales which are physical function, restricted roles due to physical problems, pain, general health, energy / vitality, social functions, mental health and mental health with restricted roles due to emotional problems. All items are evaluated with a 5-point Likert-type scale, and higher scores indicate better quality of life.
Fear Avoidance Beliefs Questionnaire | 1 day
  The FABQ measures athletes' fear of pain and consequent avoidance of physical activity or sports because of their increased fear. The questionnaire contains 16 items between 0 and 6 while 0 indicates completely disagree and 6 indicates completely agree. The maximum score is 96 and higher scores indicates increased level of fear avoidance beliefs.

CONTACTS AND LOCATIONS:
Locations (1):
- Sportomed Fulya Physiotherapy Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No